CLINICAL TRIAL: NCT03558165
Title: Lung Cancer Next Generation Sequencing Using the Oncomine Comprehensive Cancer Panel
Brief Title: Lung Cancer Next Generation Sequencing Using the Oncomine Comprehensive Assay
Acronym: LU-NGS-2
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); The Princess Margaret Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 17-5638
Record Dates: First submitted 2018-05-07; First posted 2018-06-15 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage IV Lung Adenocarcinoma
  Interventions: Diagnostic Test: Oncomine Comprehensive Assay

INTERVENTIONS:
Diagnostic Test: Oncomine Comprehensive Assay — Stage IV lung adenocarcinoma patients will have previously biopsied tumor tissue tested with the Oncomine Comprehensive Assay

SUMMARY:
Currently, publicly funded standard of care testing in Ontario for stage IV lung cancer patients uses individual gene tests to look for mutations in the EGFR and ALK genes. This testing broadens treatment options for patients, however there are other gene mutations with corresponding targeted treatments that are not routinely tested for. This study will evaluate the utility and added value of using a next generation sequencing (NGS) panel, the Oncomine Comprehensive Assay v3, to profile stage IV lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Pathologic or cytologic confirmation of lung adenocarcinoma (mixed adenocarcinoma and sarcomatoid features permitted)
* Stage IV disease
* Sufficient FFPE tumour tissue for OCCP testing
* Performance status 0-2
* Candidates for targeted therapy (TKIs) and/or clinical trials as determined by the patient's medical oncologist
* Prognosis > 6 months
* Known translocations of RET, MET exon14 skipping variants, or MET amplification are allowed

Exclusion Criteria:

● Patients with known EGFR, KRAS, BRAF and ERBB2 mutations or ALK or ROS1 fusions at study entry unless acquired resistance to molecularly targeted therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be recruited at outpatient thoracic oncology clinics at the Princess Margaret Cancer Centre.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2022-02-18 (Actual)

PRIMARY OUTCOMES:
Incremental actionable targets | 8-12 weeks from Oncomine Comprehensive Assay testing
  Calculate the number of incremental actionable targets identified by the Oncomine Comprehensive Assay compared to current standard of care molecular profiling (EGFR, ALK) in patients with stage IV NSCLC.
Number of clinical trial opportunities | 1 year from Oncomine Comprehensive Assay testing
  Compile the number of clinical trial opportunities that patients with stage IV NSCLC would be eligible for based on targets identified by the Oncomine Comprehensive Assay compared to standard of care molecular profiling (EGFR, ALK).

SECONDARY OUTCOMES:
Test turnaround time | To be assessed after accruing 50 patients (up to 2.5 years) and after 100 patients (up to 5 years).
  Calculate the time to receive Oncomine Comprehensive Assay results compared to the standard of care tissue molecular test turnaround time (EGFR, ALK).
Financial feasibility | To be assessed after accruing 50 patients (up to 2.5 years) and after 100 patients (up to 5 years).
  Perform a cost consequence analysis to evaluate financial feasibility of the Oncomine Comprehensive Assay.
Patient willingness-to-pay | To be assessed after accruing 50 patients (up to 2.5 years) and after 100 patients (up to 5 years).
  Evaluate patient willingness-to-pay for using a next generation sequencing assay, like the Oncomine Comprehensive Assay, using a validated patient survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Perdrizet K, Stockley TL, Law JH, Smith A, Zhang T, Fernandes R, Shabir M, Sabatini P, Youssef NA, Ishu C, Li JJ, Tsao MS, Pal P, Cabanero M, Schwock J, Ko HM, Boerner S, Ruff H, Shepherd FA, Bradbury PA, Liu G, Sacher AG, Leighl NB. Integrating comprehensive genomic sequencing of non-small cell lung cancer into a public healthcare system. Cancer Treat Res Commun. 2022;31:100534. doi: 10.1016/j.ctarc.2022.100534. Epub 2022 Feb 18. PMID 35278845